CLINICAL TRIAL: NCT05138094
Title: LIVACOR Trial: Minimally Invasive LIVer And Simultaneous COlorectal Resection
Acronym: LIVACOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Hospital Southampton NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); King's College Hospital NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Plymouth NHS Trust (Other); Mauriziano Umberto I Hospital (Other); University Hospital Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); San Raffaele University Hospital, Italy (Other); Ospedali Riuniti Ancona (Other); Azienda Usl di Bologna (Other Government); Azienda Ospedaliero-Universitaria di Modena (Other); Federico II University (Other); Parma University Hospital (Other); Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie (Other); Maastricht University Medical Center (Other); University of Navarrra Hospital (Clinica Universitaria) (Other); Hospital del Mar (Other); Assistance Publique - Hôpitaux de Paris (Other); Oslo University Hospital (Other); Ziekenhuis Oost-Limburg (Other); General Hospital Groeninge (Other); Moscow Clinical Scientific Center (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP3969
Record Dates: First submitted 2021-11-05; First posted 2021-11-30 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Neoplasms Malignant; Neoplasm Metastasis
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive two-stage resection (Active Comparator): Minimally invasive resection of the primary colorectal carcinoma and liver metastases in two stages. The liver metastases or the colorectal carcinoma can be resected during the first surgical procedure.
  Interventions: Procedure: Minimally invasive two-stage resection
- Minimally invasive simultaneous resection (Experimental): Minimally invasive resection of both the primary colorectal carcinoma and the liver metastases in one procedure.
  Interventions: Procedure: Minimally invasive simultaneous resection

INTERVENTIONS:
Procedure: Minimally invasive simultaneous resection — One minimally invasive surgical procedure wherein both the primary colorectal carcinoma and the liver metastases are removed.
  Other Names: Minimally invasive combined resection; Minimally invasive synchronous resection
  Arms: Minimally invasive simultaneous resection
Procedure: Minimally invasive two-stage resection — Two minimally invasive surgical procedures wherein the primary colorectal carcinoma and the liver metastases are removed
  Other Names: Minimally invasive sequential resection
  Arms: Minimally invasive two-stage resection

SUMMARY:
The LIVACOR - Trial is a European wide, randomized controlled, open-label, multicenter trial. Patients with synchronous colorectal liver metastases (CRLMs) and primary colorectal tumor are considered eligible and will be randomized between minimally invasive (MI) combined or staged colorectal resection (all colectomies, including high anterior resection) and liver resection of up to three segments.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Diagnosed with primary CRC with resectable synchronous CRLMs (with or without neoadjuvant chemotherapy)*
* Elective indication for MI combined or staged colorectal resection (all colectomies, including high anterior resection) and liver resection of up to 3 segments with a maximum of 2 separate liver resections. The MI two-staged approach includes both the conventional strategy (first resection of primary colorectal tumor followed by liver resection for CRLMs) and liver-first strategy (first CRLMs resection followed by resection of colorectal primary tumor). Patients undergoing bilobar resections are eligible (if 3 or fewer segments are resected)
* BMI between and including 18-35
* Patients with American Society of Anesthesiologists (ASA) physical status I-III and the American College of Surgeons national surgical quality improvement project (ACS NSQIP) universal surgical risk score of ≤ 50% for serious complications

  * In case of neoadjuvant chemotherapy, time interval between last chemotherapy cycle and (first) surgery should be 4-6 weeks.

Exclusion Criteria:

* Inability to give (written) informed consent.
* Patients requiring a planned temporarily or permanent stoma after colorectal resection (all colectomies, including high anterior resection). Patients who will receive an unplanned stoma intraoperatively, will be analysed according to their initial treatment assignment.
* Patients requiring multivisceral colorectal resection (all colectomies, including high anterior resection).
* Indication for MI combined or staged low anterior resection, total mesorectal excision or abdominoperineal resection and liver resection of four or more segments (i.e., hemihepatectomy or more extensive resections).
* Patients with peritoneal metastases.
* Patients with ASA physical status IV-V and ACS NSQIP surgical risk score of > 50% for serious complications.
* Repeat open hepatectomy
* Surgical history of colorectal- or liver resection for neoplastic disease
* Surgical history of major or complicated open abdominal surgery
* Indication for concurrent thermal ablation
* Medical history of thermal ablation of liver for malignancy
* Unresectable extrahepatic metastases
* Pre-operatively reconstruction of vessels/bile ducts is deemed necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to functional recovery | Expected average of 4 to 12 days postoperatively
  A patient is considered functionally recovered from a surgical procedure when several pre-specified criteria have been met.

SECONDARY OUTCOMES:
R0 resection margin | 30 days postoperatively
  Proportion of patients in whom a microscopically radical resection of both the primary colorectal carcinoma and the liver metastases was performed.
Length of hospital stay | 30 days postoperatively
  The length of hospital stay for the surgical procedure(s)
Activity tracking using Fitbit™ | 14 days pre-operatively and 60 days postoperatively
  A patient's functional recovery will also be assessed using the Fitbit smartwatch.
Intraoperative blood loss | During the surgical procedure
  Intraoperative blood loss in milliliters
Operative time | Operative time from incision until last suture
  Operative time in minutes
Morbidity | 90-days postoperatively
  Morbidity related to the surgical procedure(s)
Postoperative bile leakage | 90-days postoperatively
  Bile leakage occurring after the liver resection
Postoperative anastomotic leakage | 90-days postoperatively
  Anastomotic leakage occurring after the colorectal resection
Conversion to open surgery | During the surgical procedure
  Intra-operative conversion to an open or hand-assisted procedure
Readmission rate | 90-days postoperatively
  Proportion of patients who is unexpectedly readmitted after the surgical procedure(s)
Health-Related Quality of Life | 1 year postoperatively
  The physical, social and emotional well-being of the patient; assessed using the EuroQol 5d and European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 instruments.
Reasons for delay of discharge after functional recovery | 30 days postoperatively
  All reasons that may cause delay in discharge after the patient has recovered functionally, such as administrative reasons, patient confidence, logistics problems, etc.
Hospital and societal costs | 1 year postoperatively
  All costs that are associated with the operation, including in-hospital costs and out of hospital costs, such as home care, work absence, etc.
Three and five-year recurrence free survival | 5 years postoperatively
  The proportion of patients which is free of recurrence of the malignant disease after resection of both the primary colorectal carcinoma and the liver metastases.
Three and five-year overall survival | 5 years postoperatively
  The proportion of patients which is alive after resection of both the primary colorectal carcinoma and the liver metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Mohammed Abu Hilal, MD PhD, Study Chair — Fondazione Poliambulanza Istituto Ospedaliero
Locations (28):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - General Hospital Groeninge, Kortrijk, West Flanders
- Antoine-Béclère Hospital, Paris, Île-de-France Region, France
- Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie, Saarbrücken, Saarland, Germany
- Italy (10):
  - Federico II University Hospital, Naples, Calabria
  - Azienda USL di Bologna, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Modena, Modena, Emilia-Romagna
  - Parma University Hospital, Parma, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Lombardy
  - San Raffaele University Hospital, Milan, Lombardy
  - Mauriziano Umberto I Hospital, Turin, Piedmont
  - Ospedali Riuniti, Ancona, The Marches
  - University Hospital Padova, Padua, Veneto
- Centre Hospitalier du Luxembourg, Luxembourg, Luxembourg
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Amsterdam UMC, Amsterdam, North Holland
- Oslo University Hospital, Oslo, Østlandet, Norway
- Moscow Clinical Scientific Center, Moscow, Moscow Oblast, Russia
- Spain (2):
  - Hospital del Mar, Barcelona, Catalonia
  - University of Navarrra Hospital (Clinica Universitaria), Pamplona, Navarre
- United Kingdom (7):
  - Manchester University NHS Foundation Trust, Manchester, North West England
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle, Northeast England
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, Northwest England
  - University Hospital Southampton NHS Foundation Trust, Southampton, South East England
  - King's College Hospital NHS Trust, London, Southeast England
  - University Hospital Plymouth NHS Trust, Plymouth, Southwest England
  - University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Poel MJ, Tanis PJ, Marsman HA, Rijken AM, Gertsen EC, Ovaere S, Gerhards MF, Besselink MG, D'Hondt M, Gobardhan PD. Laparoscopic combined resection of liver metastases and colorectal cancer: a multicenter, case-matched study using propensity scores. Surg Endosc. 2019 Apr;33(4):1124-1130. doi: 10.1007/s00464-018-6371-1. Epub 2018 Aug 1. PMID 30069639
- [Background] Pan L, Tong C, Fu S, Fang J, Gu Q, Wang S, Jiang Z, Juengpanich S, Cai X. Laparoscopic procedure is associated with lower morbidity for simultaneous resection of colorectal cancer and liver metastases: an updated meta-analysis. World J Surg Oncol. 2020 Sep 21;18(1):251. doi: 10.1186/s12957-020-02018-z. PMID 32958079
- [Background] Boudjema K, Locher C, Sabbagh C, Ortega-Deballon P, Heyd B, Bachellier P, Metairie S, Paye F, Bourlier P, Adam R, Merdrignac A, Tual C, Le Pabic E, Sulpice L, Meunier B, Regimbeau JM, Bellissant E; METASYNC Study group. Simultaneous Versus Delayed Resection for Initially Resectable Synchronous Colorectal Cancer Liver Metastases: A Prospective, Open-label, Randomized, Controlled Trial. Ann Surg. 2021 Jan 1;273(1):49-56. doi: 10.1097/SLA.0000000000003848. PMID 32209911
- [Background] Gavriilidis P, Sutcliffe RP, Hodson J, Marudanayagam R, Isaac J, Azoulay D, Roberts KJ. Simultaneous versus delayed hepatectomy for synchronous colorectal liver metastases: a systematic review and meta-analysis. HPB (Oxford). 2018 Jan;20(1):11-19. doi: 10.1016/j.hpb.2017.08.008. Epub 2017 Sep 7. PMID 28888775